CLINICAL TRIAL: NCT03419806
Title: Levodopa Pharmacokinetics in Patients With Parkinson's Disease and Symptom Fluctuation: A Phase I, Open-label, Randomized, Multicentre, Crossover Study Comparing Intravenous and Subcutaneous Infudopa With Intestinal Duodopa
Brief Title: Study Comparing Intravenous and Subcutaneous Infudopa With Intestinal Duodopa in Patients With Parkinson's Disease
Acronym: IPO-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: The Swedish Research Council (Other Government); Dizlin Medical Design AB (Unknown); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-002488-17
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Infudopa i.v. (Experimental): Infudopa i.v. in 75% of the subject's individual pre-study dosing of Duodopa will be delivered over a 16-h period, administered as a morning rapid i.v. constant rate administration followed by continuous i.v. infusion.
  From patient 6 and onwards:
  Infudopa i.v. in 81% of the subject's individual pre-study dosing of Duodopa will be delivered over a 16-h period, administered as a morning rapid i.v. constant rate administration followed by continuous i.v. infusion.
  Interventions: Drug: Infudopa i.v.
- Infudopa s.c. (Experimental): Infudopa s.c. in the same dosage as the subject's individual pre-study dosing of Duodopa will be delivered over a 16-h period, administered as a morning rapid s.c. constant rate administration followed by continuous s.c. infusion.
  From patient 6 and onwards:
  Infudopa s.c. in 86% of the subject's individual pre-study dosing of Duodopa will be delivered over a 16-h period, administered as a morning rapid s.c. constant rate administration followed by continuous s.c. infusion.
  Interventions: Drug: Infudopa s.c.
- LCIG (Duodopa) (Active Comparator): Individually optimized dosing of LCIG (Duodopa) (delivered directly to the proximal small intestine via a percutaneous endoscopic gastrojejunostomy (PEG-J) tube connected to a portable infusion pump) will be delivered over a 16-h period, administered as a morning rapid constant rate administration followed by continuous infusion.
  Interventions: Drug: LCIG (Duodopa)

INTERVENTIONS:
Drug: Infudopa i.v. — Infudopa i.v. infusion will be given through an indwelling catheter placed in the arm. Infudopa i.v. will be delivered in 75% of the subject's individual pre-study dosing of Duodopa.
  From patient 6 and onwards:
  Infudopa IntraV, at 81% of the subject's individual pre-study daily Duodopa dose, will be delivered over a 16-h period and administered as a continuous fixed infusion rate preceded by a morning bolus dose. The i.v. morning bolus is 110% of the hourly continuous dose delivered at the rate of 60 ml/h (mixed volume rate Infudopa Active + Infudopa Buffer IntraV). The morning dose will not exceed 24 mL, corresponding to 240 mg levodopa. The maximum daily dose levodopa during i.v. administration is not allowed to exceed 3240mg (equal to 81% of the maximum allowed daily dosage for Duodopa that is 4000 mg).
  Other Names: Infudopa IntraV
  Arms: Infudopa i.v.
Drug: Infudopa s.c. — A suitable infusion needle will be placed laterally on the abdomen for the s.c. infusion of Infudopa. Infudopa s.c. will be delivered in the same dosage as the subject's individual pre-study dosing of Duodopa, as a morning rapid s.c. constant rate administration followed by continuous s.c. infusion up to 16 h.
  From patient 6 and onwards:
  Two infusion needles will be placed on the abdomen for the s.c. infusion of Infudopa SubC in 86% of the the subject's individual pre-study daily Duodopa dose. The intervention is given as a continuous fixed infusion rate for 16h preceded by a morning bolus dose. The s.c. morning bolus is 155% of the hourly continuous dose delivered at the rate of 80 ml/h (mixed volume rate Infudopa Active + Infudopa Buffer SubC). The morning dose will not exceed 30 mL. The maximum daily dose levodopa during s.c. administration is not allowed to exceed 3440mg (equal to 86% of the maximum allowed daily dosage for Duodopa that is 4000 mg).
  Other Names: Infudopa SubC
  Arms: Infudopa s.c.
Drug: LCIG (Duodopa) — Duodopa will be administered directly to the proximal small intestine via a PEG-J tube connected to a portable infusion pump. Individually optimized dosing of Duodopa will be administered as a morning rapid constant rate administration followed by continuous infusion and, if needed, intermittent extra doses (subject-initiated based on symptom experience). The maximum daily dose levodopa during Duodopa administration should normally not exceed 3350 mg, and is not allowed to exceed 4000 mg.
  From patient 6 and onwards:
  The pre-study daily Duodopa dose will be delivered over a 16-h period and administered as a continuous fixed infusion rate preceded by a morning bolus dose. The morning bolus is 110% of the hourly continuous dose delivered at the rate of 40 ml/h. The morning dose will not exceed 15 mL, corresponding to 300 mg levodopa. The maximum daily dose levodopa is not allowed to exceed 4000mg.
  Arms: LCIG (Duodopa)

SUMMARY:
In patients with Parkinson's disease, the characteristic motor symptoms, i.e., slowness of movement (bradykinesia), tremor and rigidity, are consequences of the progressive degeneration of neurons containing and releasing dopamine. The first-line treatment of Parkinson´s is oral administration of levodopa - a precursor to dopamine that (unlike dopamine) passes the blood brain barrier. After the first few years of treatment with levodopa, many patients do however develop a highly variable response to the drug characterised by rapid shifts between impaired locomotion and drug induced dyskinesias (referred to as the on-off syndrome). This is cased by the marked variation in serum levodopa levels following per oral administration, and it is known that intravenous administration of levodopa give a more stable level of levodopa with improved on-off symptoms.

Levodopa-carbidopa intestinal gel (LCIG) - under the name of Duodopa® - is delivered directly to the proximal jejunum via a tube connected to a portable infusion pump. Infusion of Duodopa in the jejunum bypasses gastric emptying, helping to avoid the fluctuation in plasma levodopa levels. However, while clearly confirming that an even administration of levodopa is of considerable benefit to Parkinson patients with on-off symptomatology, the LCIG approach is marred by the need for surgery (for the insertion of the intestinal tube) and various possible complications following this, as well as by side effects such as abdominal pain.

Researchers have now succeeded in producing a physiologically acceptable levodopa solution (called Infudopa) in a concentration allowing for a continuous intravenous (i.v.) or subcutaneous (s.c.) administration of therapeutic doses to humans. Early experience of this strategy confirms that both s.c. and i.v. administration of this solution results in even serum levodopa levels and markedly improved motor functioning. The aim of this study is to compare the pharmacokinetic profile of Infudopa administered i.v. and s.c. with that of Duodopa administered enterally in parkinsonian patients with on-off complications.

DETAILED DESCRIPTION:
IPO-001 is a prospective, randomized, 3-period cross-over, open-label multicentre trial comparing intravenous and subcutaneous Infudopa with intestinal Duodopa. The patients will be identified and recruited at neurology clinics at university hospital clinical sites in Sweden, and travel from their living location to a clinical phase I site with full Good Clinical Practice (GCP) standard at the Sahlgrenska University Hospital in Gothenburg for the three treatment visits.

At the phase I study clinic, patients will receive Duodopa at optimal dosage for 16 hours at one of the treatment visits, i.v. Infudopa at a concentration estimated to yield corresponding serum levels of levodopa for the same duration at another treatment visit, and they will again receive the corresponding amount of levodopa but in the form of s.c. Infudopa at a third visit. The study will hence have a cross-over design with a minimum of three days on Duodopa between the different treatment visits, where the order of treatments will be non-blinded but randomized.

Blood samples will be drawn according to a set schedule during the treatment visits, and subjects will be monitored for safety throughout the study, with focus on the local tolerability at the injection sites of i.v. and s.c. administration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male or female patients at least 30 years old
3. Patients with advanced Parkinson's disease who are already on LCIG (Duodopa®) for at least 30 days, on a stable treatment regimen of 685 mg to 4000 mg levodopa per day, and with approximately 16- or 24-h Duodopa infusion regimens*
4. Patients with a Hoehn and Yahr (H&Y) score of ≤ 3 on Duodopa treatment (including concomitant medication)
5. Body mass index range from 18.0 to 35.0 kg/m2
6. Patients in general good health, as judged by the Investigator, and as determined by vital signs, medical history, physical examination, ECG, and laboratory tests
7. Females of childbearing potential must have a negative pregnancy test prior to randomization and must be willing to use a highly effective contraceptive measure during relevant systemic exposure to the investigational drug and the first menstrual cycle after treatment cessation (see section 7.3).
8. Males must be willing to refrain from fathering a child, including sperm donation, during the study and 3 months following the last dose.

   * Criterion 3 updated to "...a stable treatment regimen of 600 mg to 4000 mg levodopa per day" after first interim analysis (patient 6 and onwards)

Exclusion Criteria**:

1. Simultaneous participation in any other clinical study 2. Known drug abuse of any kind, or other condition that may render the patient more likely to be non-compliant to the protocol, as judged by the investigator 3. Patients who are considered to be violent or patients considered at suicidal risk by the investigator 4. Clinically significant abnormal laboratory data at baseline or any abnormal laboratory value that could interfere with the study assessments 5. Patients with serious symptomatic cerebral disease, cerebrovascular disease, focal neurological lesions (previous brain surgery), any acute brain trauma requiring treatment with anticonvulsant therapy, or acute stroke 6. Current diagnosis or history of drug or alcohol abuse within 12 months of baseline 7. Other psychiatric, neurological, or behavioral disorders that may interfere with the conduct or interpretation of the study, as judged by the Investigator 8. History of, or current, seizure disorders and patients requiring treatment with anticonvulsants 9. History or presence of any condition that might interfere with absorption, distribution, metabolism, or excretion of study drug, however, the PEG/J (percutaneous endoscopic gastrojejunostomy) tube that Duodopa patients have is not considered as such condition 10. Patients on medication with warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, monoamine oxidase-A inhibitors and alpha-methyldopa (within last 60 days); selegiline, catechol-O-methyltransferase (COMT) inhibitors, dopamine, parenteral ergots, methylphenidate, amphetamine, beta blockers for treating tremor, isoprenaline, adrenaline, dobutamide, reserpine, flunarizine or cinnarizine, isoniazid, metoclopramide, and anticholinergics (within last 30 days); and iron salts (within last 7 days), or any other treatment that could affect the metabolism of levodopa 11. Patients who use antineoplastic and immunosuppressants (within the last 5 years), and drugs known to increase risks for cardiac toxicity, Torsade de Pointes, sudden death or prolonged QT interval (within five elimination half-lives before baseline and for the duration of the study)

**) Replaced by the following exclusion criteria after interim analysis (patient 6 and onwards):

1. Simultaneous participation in any other clinical drug trial
2. Clinically significant abnormal laboratory data at baseline or any abnormal laboratory value that could interfere with the study assessments.
3. Patients with current serious symptomatic CNS-lesions, neurological, psychiatric, or behavioral disorders other than Parkinson's disease (e.g. major stroke, epilepsy, substance use disorder, previous neurosurgery including DBS) and that may interfere with the conduct or interpretation of the study
4. History or presence of any condition that can interfere with absorption, distribution, metabolism, or excretion of study drug (not including the percutaneous endoscopic gastrojejunostomy tube needed for Duodopa administration)
5. Patients on medication with warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, monoamine oxidase-A inhibitors and alpha-methyldopa (within the last 60 days); selegiline, catechol-O-methyltransferase (COMT) inhibitors other than a single daily dose of entacaponeparenteral ergots, anticholinergics, methylphenidate, amphetamine, isoprenaline, adrenaline, dobutamide, reserpine, or other drugs with known dopamine receptor antagonistic effect (within the last 30 days); and iron salts (within the last 7 days), or any other treatment that could affect the metabolism of levodopa
6. Patients who use antineoplastic chemotherapy or biological immunosuppressants (within the last 5 years), and drugs known to increase risks for cardiac toxicity, Torsade de Pointes, sudden death or prolonged QT interval (within five elimination half-lives before baseline and for the duration of the study)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentration - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  To demonstrate that Infudopa i.v. and s.c. yield steady state plasma concentration of levodopa that is equivalent with that of Duodopa.
Area under plasma concentration versus time curve (AUC) - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  AUC of levodopa plasma concentrations during the dosage interval with Infudopa i.v. and s.c. will be compared to Duodopa.
Coefficient of variation (COV) for plasma levodopa concentrations | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  COV for plasma levodopa concentrations during the dosage interval with Infudopa i.v. and s.c. will be compared to Duodopa.

SECONDARY OUTCOMES:
Local skin tolerability to the investigated products, Draize score | For each treatment visit - Baseline: Day -1; Post infusion: t=24h, day 30±5 (only s.c. infusion), 30+/-5 days after last treatment visit.
  The number of participants with treatment-related local skin reactions during or following s.c and i.v. infusion of the IMP will be assessed. Local skin reactions will be rated by a dermatologist using Draize scoring.
Local skin tolerability to the investigated products, subjective symptom ratings | For each treatment visit: Day 1 during infusion: t=2h, t=8h, t=16h after infusion start; Day 2 post infusion: t=24h after infusion start, day 30±5 (only s.c. infusion), 30+/-5 days after last treatment visit.
  In participants with skin reactions the skin symptoms tenderness and itching will be rated by the participants using a horizontal 10 cm visual analogue scale graded 0-100 where 0 represents no symptom and 100 worst possible.
Bioavailability - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  To establish the bioavailability of levodopa given s.c. and as Duodopa compared to the i.v. administration
Bioavailability - carbidopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  To establish the bioavailability of carbidopa given s.c. and as Duodopa compared to the i.v. administration
Maximum plasma concentration (Cmax) - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare maximum plasma concentration (Cmax) of levodopa during treatment with s.c and i.v Infudopa versus Duodopa.
Maximum plasma concentration (Cmax) - carbidopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare maximum plasma concentration (Cmax) of carbidopa during treatment with s.c and i.v Infudopa versus Duodopa.
Time of the maximum plasma concentration (tmax) - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare time of the maximum plasma concentration (tmax) of levodopa during treatment with s.c and i.v Infudopa versus Duodopa.
Time of the maximum plasma concentration (tmax) - carbidopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare time of the maximum plasma concentration (tmax) of carbidopa during treatment with s.c and i.v Infudopa versus Duodopa.
Area under the curve (AUC) - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare area under the curve (AUC) of levodopa during treatment with s.c and i.v Infudopa versus Duodopa.
Area under the curve (AUC) - carbidopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare area under the curve (AUC) of carbidopa during treatment with s.c and i.v Infudopa versus Duodopa.
Elimination half-life (t½) - levodopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare elimination half-life (t½) of levodopa during treatment with s.c and i.v Infudopa versus Duodopa.
Elimination half-life (t½) - carbidopa | For each treatment visit: Pre-dose, t=15 min, t=30 min, t=1h, t=1.5h, t=2h, t=2.5h, t=3h, t=3.5h, t=4h, t=5h, t=6h, t=7h, t=8h, t=10h, t=12h, t=14h, t=16h, t=16.5h, t=17h, t=17.5h, t=18h, t=23h, and t=24h from infusion start.
  Compare elimination half-life (t½) of carbidopa during treatment with s.c and i.v Infudopa versus Duodopa.
Parkinson's disease motor symptom ratings | For each treatment visit: pre-dose, t=1,5h, t=5h, t=6h, t=7h, t=16h and t=24h from infusion start.
  Bradykinesia and dyskinesia will be assessed using the Treatment Response Scale, TRS (Nyholm et al, 2005). For this assessment the following items from the UPDRS will be performed: Finger tapping (item 23), Rapid alternating hand movements (item 25), eg agility (item 26), arising from chair (item 27), gait (item 29), and global bradykinesia (item 31). The occurrence of dyskinesia during these items will be assessed according to the definitions of the Modified Dyskinesia Scale (Goetz et al. 1994). The TRS outcome measure is a Likert scale that ranges from -3 to +3 (severely bradykinetic to severely dyskinetic).
Parkinson Kinetigraph objective bradykinesia measurement (BK score) | For each treatment visit: Between 9-18 as well as +1h to +16h after infusion start.
  The 25th, 50th and 75th percentiles of the BK scores from a 24h recording will be determined.
Parkinson Kinetigraph objective dyskinesia measurement (DK score) | For each treatment visit: Day 1: Between 9-18 as well as +1h to +16h after infusion start.
  The 25th, 50th and 75th percentiles of the DK scores from a 24h recording will be determined.
Parkinson Kinetigraph objective tremor episodes | For each treatment visit: Day 1: Between 9-18 as well as +1h to +16h after infusion start.
  The percent of time with ongoing tremor consisting of at least 10 seconds meeting the operational tremor criteria defined by Braybrook et al (2016) will be measured.
Parkinson Kinetigraph objective Fluctuation dyskinesia score (FDS) | For each treatment visit: Day 1: Between 9-18 as well as +1h to +16h after infusion start.
  The fluctuation dyskinesia score will be calculated from the interquartile range of BK and DK scores.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Bergquist, Ass Prof, Principal Investigator — Department of Pharmacolgy at Institute of Neuroscience and Physiology
Locations (1):
- Sahlgrenska Universtiy Hospital, Dep of Neurology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergquist F, Ehrnebo M, Nyholm D, Johansson A, Lundin F, Odin P, Svenningsson P, Hansson F, Bring L, Eriksson E, Dizdar N. Pharmacokinetics of Intravenously (DIZ101), Subcutaneously (DIZ102), and Intestinally (LCIG) Infused Levodopa in Advanced Parkinson Disease. Neurology. 2022 Sep 5;99(10):e965-e976. doi: 10.1212/WNL.0000000000200804. PMID 35705502